CLINICAL TRIAL: NCT01071785
Title: Dietetic Intervention With Soluble Fiber in Type 2 Diabetes Mellitus (DM) Patients With Metabolic Syndrome (MS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Mirela jobim de Azevedo, Federal University of Rio GRAnde do sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCPA-06370
Record Dates: First submitted 2008-06-06; First posted 2010-02-19 (Estimated); Last update posted 2010-03-01 (Estimated); Status verified 2010-02

CONDITIONS: Metabolic Syndrome; Albuminuria
Keywords: Metabolic Syndrome; diet; fiber; Serum lipids; Albuminuria
MeSH Terms: conditions — Metabolic Syndrome; Albuminuria | interventions — guar gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual diet (No Intervention): no dietary or drug intervention. Patients followed their usual diet.
- guar gum (Experimental): guar gum
  Interventions: Dietary Supplement: guar gum

INTERVENTIONS:
Dietary Supplement: guar gum — guar gum 10g/day for six weeks
  Other Names: benefiber; guar gum group
  Arms: guar gum

SUMMARY:
Metabolic Syndrome (MS) is an clinical condition with high cardiovascular risk. More than 80% of DM patients had MS. Dietary factors can be associated to both, DM and MS. Therefore the aim of this study is to evaluate the effects of add soluble fiber (goma-guar) in the usual diet of type 2 DM with MS and compare this intervention with an usual diet without this supplement.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effect of soluble fiber (guar gum) on the MS components (International Diabetes Federation-2005 and WHO): blood pressure, plasma glucose, triglycerides, HDL, central obesity (waist, BMI),and albuminuria. Secondary objectives are: effect of guar gum on serum fatty acids, , PCR, endothelin 1, and fibrinogen. Primary outcomes were alterations on MS components.

Forty-four type 2 diabetic outpatients were included in a randomized clinical trial: treatment 1- guar gum (10g/day) + usual diet; treatment 2- usual diet. The duration of each treatment was six weeks. Three days weight diet records with concurrent 24h urinary collections (protein intake estimative), clinical and laboratory evaluation were performed at baseline and after 4 and 6 weeks. Serum fatty acids were measured in total triglycerides fractions by gas chromatography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Using metformin and/or Insulin

Exclusion Criteria:

* serum triglycerides > 400 mg/dl
* serum creatinine > 2 mg/dl
* gastrointestinal malabsorption

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Changes on the components of metabolic syndrome (according to IDF and WHO criteria): blood pressure, waist, body mass index (BMI), triglycerides, high-density lipoprotein (HDL) cholesterol, glucose values (HBA1c) and urinary albumin excretion. | 4 and 6 weeks

SECONDARY OUTCOMES:
changes on serum fatty acids and serum cholesterol | 4 and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mirela J Azevedo, MD, Principal Investigator — HCPA; Jorge L Gross, MD, Study Director — HCPA; Valesca Dall'Alba, RD, Principal Investigator — HCPA
Locations (1):
- HCPA, Porto Alegre, Rio Grande do Sul, Brazil